CLINICAL TRIAL: NCT03815500
Title: Patient Education at Dismissal After Surgical Procedure: Clinical Outcome Implications and Improvement Strategies
Brief Title: Patient Education at Dismissal After Surgical Procedure
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI no longer with the organization, no subjects enrolled
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 18-008124
Record Dates: First submitted 2019-01-08; First posted 2019-01-24 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: Wound Infection Post-Traumatic; Wound Infection; Wound Complication; Wound Breakdown; Wound Open
MeSH Terms: conditions — Wound Infection; Surgical Wound Dehiscence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with open surgical wounds (Experimental): Patients with open surgical wounds will undergo enhanced packing education with curriculum designed for learners with low literacy, dyslexia or associated learning disorders.
  Interventions: Behavioral: Enhanced Education

INTERVENTIONS:
Behavioral: Enhanced Education — Enhanced educational curriculum will involve learning modalities including 3D modeling, video, and visual-aid enhanced text for references to improve caregiver and patient understanding of wound packing techniques.

SUMMARY:
Can improvements in patient dismissal education materials reduce incidence of wound non-healing and infection.

DETAILED DESCRIPTION:
The investigators seek to address the specific educational needs of patients and caregivers with low-literacy, dyslexia and related learning disabilities in the context of properly performing wound care for patients with surgical wounds. Specific aims include both improving care by decreasing wound complications and improving patient satisfaction by using techniques designed for this population. Objectives include utilizing surveys to determine the incidence of dyslexia among the patients' and caregivers' within the general surgery service as well as the perception of our current educational offerings, to design a new dismissal package with enhanced educational offerings, to re-measure this effect on the patient experience with survey data, and to compare wound infection rates before and after implementing the new curriculum. Dyslexia and associated learning disabilities are common and likely impact the health literacy among this population due to the ubiquitous literacy-based documentation of hospital course and dismissal instructions. Adults with dyslexia may be reluctant to disclose any inability to understand written instructions. There is currently no mechanism within the dismissal system to specifically identify and address the unique needs of this population. The impact on clinical outcomes of proper wound packing is substantial, and if performed incorrectly can lead to slow wound healing and infections that often require readmission, multiple courses of antibiotics, and reoperation. In severe cases, improper wound care can lead to severe infection, sepsis, and death. By enhancing the educational offerings of proper wound care to this population, the investigators hope to reduce these complications.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients on the general surgery service with open wounds requiring packing

Exclusion Criteria:

* Patients with wound vacs
* Patients receiving exclusively professional wound care or home health services

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Utilization of education curriculum designed for learners with low literacy, dyslexia and associate learning disorders | 6 months
  Nursing surveys answering the question, "Have you been trained to teach wound care to patients with dyslexia or learning disabilities?" Were answered "No," by 43/46 (93%) respondents. We seek to have a 90% rate of affirmative ("Yes") answers to this survey after implementation of our curriculum.

SECONDARY OUTCOMES:
Patient satisfaction with wound education | 6 months
  Survey of patients' wound education experiences should indicate that they are being offered curriculum suitable for learners with low literacy, dyslexia and associated learning disorders. We will utilize a scale of "Definitely satisfied, somewhat satisfied, somewhat dissatisfied, definitely dissatisfied" as our measure.
shorter time to wound healing | 1 year
  After implementation of new curriculum, it is anticipated that wound complication rates and time to wound healing would decrease. We will calculate the "time" based on the date of wound creation to their final clinic appointment indicated the wound is satisfactorily healed with "days" as our unit of measure.

CONTACTS AND LOCATIONS:
Overall Officials: Martin D Zielinski, Principal Investigator — Mayo Clinic

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials